CLINICAL TRIAL: NCT00006348
Title: Phase III, Randomized, Double-Blind, Placebo-Controlled Crossover Trial of Ondansetron in the Control of Chronic Nausea and Vomiting Not Due to Antineoplastic Therapy in Patients With Advanced Cancer
Brief Title: Ondansetron in Treating Patients With Advanced Cancer and Chronic Nausea and Vomiting Not Caused by Cancer Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-989201; CDR0000068205 (Registry Identifier: PDQ (Physician Data Query)); NCI-P00-0168
Record Dates: First submitted 2000-10-04; First posted 2004-03-25 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Nausea and Vomiting; Precancerous Condition; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenström macroglobulinemia; stage III multiple myeloma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; small intestine lymphoma; unspecified childhood solid tumor, protocol specific; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated childhood acute lymphoblastic leukemia; polycythemia vera; primary myelofibrosis; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; primary central nervous system non-Hodgkin lymphoma; nausea and vomiting; prolymphocytic leukemia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; primary systemic amyloidosis; intraocular lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Nausea; Vomiting; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Recurrence; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Intraocular Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: ondansetron + placebo (Experimental): Patients receive oral ondansetron twice daily on days 1-7 and oral placebo twice daily on days 8-14 in the absence of unacceptable toxicity.
  Interventions: Drug: ondansetron; Other: placebo
- Arm 2: ondansetron + placebo (Experimental): Patients receive oral placebo twice daily on days 1-7 and oral ondansetron twice daily on days 8-14 in the absence of unacceptable toxicity.
  Interventions: Drug: ondansetron; Other: placebo

INTERVENTIONS:
Drug: ondansetron
Other: placebo

SUMMARY:
RATIONALE: Antiemetic drugs, such as ondansetron, may help to reduce or prevent nausea and vomiting in patients with advanced cancer.

PURPOSE: This randomized phase III trial is studying how well ondansetron works compared to a placebo in treating patients with advanced cancer and chronic nausea and vomiting that is not caused by cancer therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the antiemetic effect of ondansetron vs placebo in patients with advanced cancer who suffer from chronic nausea and emesis that is not due to antineoplastic therapy (i.e., chemotherapy, radiotherapy, immunotherapy, biologic therapy). II. Determine the toxicity of ondansetron in these patients. III. Evaluate the use of other concurrent antiemetics in these patients when treated with this regimen.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to abdominal carcinomatosis (yes vs no), renal insufficiency (creatinine less than 2.0 mg/dL vs creatinine at least 2.0 mg/dL), type of cancer (brain vs gastrointestinal vs other), and narcotic use (yes vs no). Patients are randomized to one of two treatment arms. Arm I: Patients receive oral ondansetron twice daily on days 1-7 and oral placebo twice daily on days 8-14 in the absence of unacceptable toxicity. Arm II: Patients receive oral placebo twice daily on days 1-7 and oral ondansetron twice daily on days 8-14 in the absence of unacceptable toxicity.

PROJECTED ACCRUAL: A total of 100 patients (50 per arm) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of incurable cancer with chronic nausea and vomiting lasting at least 1 week that is not due to antineoplastic therapy (i.e., chemotherapy, radiotherapy, immunotherapy, biologic therapy) Nausea not adequately controlled by standard antiemetics

PATIENT CHARACTERISTICS: Cardiovascular: No uncontrolled hypertension Other: Not pregnant or nursing Able to take oral medication (feeding tube allowed) Able to swallow own saliva No prior phenylketonuria No known allergy or intolerance to 5-HT3 receptor antagonists No bowel obstruction

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics At least 2 weeks since prior cytotoxic systemic therapy No concurrent cytotoxic systemic therapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 2 weeks since prior radiotherapy to gastrointestinal tract No concurrent radiotherapy to gastrointestinal tract Surgery: Not specified Other: At least 2 weeks since prior 5-HT3 receptor antagonists (i.e., dolasetron, granisetron, or ondansetron) No other concurrent 5-HT3 receptor antagonists Other concurrent antiemetics allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-10; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
response | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (12):
- United States (12):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota